CLINICAL TRIAL: NCT07317089
Title: Innovative Facial Contouring Using a Monopolar Radiofrequency Device With Continuous Water Cooling: An Integrated Clinical and Preclinical Study
Brief Title: Facial Contouring With Monopolar RF and Continuous Water Cooling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Ngoc Ha Nguyen, Principal Investigator, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIRB-23614-PM
Record Dates: First submitted 2025-12-10; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Skin Aging; Sagging Skin; Laxity; Skin
Keywords: Monopolar radiofrequency; continuous water cooling; skin rejuvenation
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm A (Experimental): Participants underwent a single RF-CWC treatment on Day 0 after eligibility screening and baseline assessments. Treatment was applied using two distinct modes based on anatomical regions. The static mode was administered to the outer facial areas, while the sliding mode was applied to the central facial areas. This approach allowed for region-specific assessment of volumetric changes corresponding to each treatment mode. Follow-up visits were conducted at weeks 2, 4, and 8.
  Interventions: Device: RF-CWC

INTERVENTIONS:
Device: RF-CWC — Participants underwent a single RF-CWC treatment on Day 0 after eligibility screening and baseline assessments. Treatment was applied using two distinct modes based on anatomical regions. The static mode was administered to the outer facial areas, while the sliding mode was applied to the central facial areas. This approach allowed for region-specific assessment of volumetric changes corresponding to each treatment mode. Follow-up visits were conducted at weeks 2, 4, and 8.

SUMMARY:
The goal of this clinical trial is to assess whether a single RF-CWC (radiofrequency - continous water cooling) session can produce significant improvements in jawline contour and facial volume in women aged 38-50 years over 8 weeks. The main questions it aims to answer are:

1. Can one session of RF-CWC elevate the jawline after 8 weeks?
2. Can one session of RF-CWC contour the lower face after 8 weeks? Researchers will compare the jawline lifting effect and mandibular volume at 2, 4, and 8 weeks to baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 38-50 years
* Agreed to abstain from any dermatological procedures, including facial lifting, during the study
* Able to adhere to the study protocol.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Failure to comply with contraception
* Facial lesions
* Hypersensitivity
* Inflammatory or infectious facial conditions
* Recent use of systemic steroids or phototherapy (within 1 month)
* Recent cosmetic procedures (within 3 months)
* Any condition deemed unsuitable by the investigator.

Ages: 38 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Jawline lifting | From baseline to the end of the study at 8 weeks
  Jawline lifting was evaluated using Morpheus3D® (Morpheus Co., Ltd., Gyeonggi, Republic of Korea), an LED-based 3D facial imaging system. Jawline lifting was measured as the curved distance (mm) from the chin to the earlobe; a decrease in length indicated improvement.
Facial volume | From baseline to the end of the study at 8 weeks
  Facial volume was evaluated using Morpheus3D® (Morpheus Co., Ltd., Gyeonggi, Republic of Korea), an LED-based 3D facial imaging system. Facial volume (ml) was assessed for two regions: the midface (between the eyes and the area from philtrum to nose), where an increase indicated volumization, and the lower face (philtrum to chin), where a decrease indicated contouring.

CONTACTS AND LOCATIONS:
Locations (1):
- Global Medical Evaluation Academy, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No